CLINICAL TRIAL: NCT04887181
Title: The Effects of Different Dentin Hypersensitivity Treatment Methods on Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kırıkkale University (Other)
Responsible Party: Principal Investigator, Behiye Esra Özdemir, Research Assistant, Kırıkkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28/02
Record Dates: First submitted 2021-05-05; First posted 2021-05-14 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Dentin Hypersensitivity
Keywords: Dentin Hypersensitivity; Desensitizing Agent; Adhesive Resin
MeSH Terms: conditions — Dentin Sensitivity | interventions — gluma desensitizer; Hybrid Bond

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teethmate Desensitizer (Active Comparator): Tetracalcium phosphate and dicalcium phosphate containing desensitizer
  Interventions: Other: Teethmate Desensitizer
- Gluma Desensitizer (Active Comparator): %35 hydroxyethyl methacrylate and %5 glutaraldehyde containing desensitizer
  Interventions: Other: Gluma Desensitizer
- Hybrid Bond (Active Comparator): Self-etch adhesive resin
  Interventions: Other: Hybrid Bond

INTERVENTIONS:
Other: Teethmate Desensitizer — Powder and liquid contained in the material were mixed. It was applied to the buccal surface of the sensitive tooth. then it was washed away from the tooth surface. 1-4 sessions were applied until the sensitivity disappeared.
  Arms: Teethmate Desensitizer
Other: Gluma Desensitizer — The material was applied to the buccal surface of the tooth with sensitivity. It was washed with water and removed from the tooth surface. 1-4 sessions were applied until the sensitivity disappeared.
  Arms: Gluma Desensitizer
Other: Hybrid Bond — It was applied to the buccal surface of the sensitive tooth with an applicator. It was cured with a LED light device. Dentin sensitivity was checked with evaporative air application. The process was repeated until the sensitivity disappeared.
  Arms: Hybrid Bond

SUMMARY:
The aim of this study was to evaluate the effects of a self etch adhesive resin and two desensitizing agents(Calcium phosphate, 5% glutaraldehyde) in treatment of dentin hypersensitivity on the quality of life of individuals.

DETAILED DESCRIPTION:
This in-vivo study was done among 69 participants who reported at least one sensitivite tooth(Schiff Sensitivity Score >1) as a result of the clinical examination. Participants were randomly divided into three treatment groups(n=23):

I. Tetracalcium phosphate and dicalcium phosphate containing desensitizer (Teethmate Desensitizer) II. %35 hydroxyethyl methacrylate and %5 glutaraldehyde containing desensitizer (Gluma Desensitizer) III. Self-etch adhesive resin (Hybrid Bond) These materials used in treatment of dentin hypersensitivity in 6 months clinical follow-up and the effects on the quality of life of individuals were evaluated with Dentine Hypersensitivity Experience Questionnaire (DHEQ).

ELIGIBILITY:
Inclusion Criteria:

* Not having any systemic disease,
* 18 years and older,
* At least one tooth complaining of dentin hypersensitivity (Schiff score> 1),
* The acceptance of the volunteers participating in the research.

Exclusion Criteria:

* Active periodontal disease,
* Periodontal surgery for the last 3 months,
* Use of desensitizing toothpaste or mouthwash in the last 3 months,
* Long-term use of analgesic and anti-inflammatory drugs,
* Having a history of allergies,
* Women during pregnancy or breastfeeding,
* Parafunctional habits (bruxism, teeth grinding etc.),
* The presence of caries, pulpitis or restoration in teeth,
* Tooth tissue loss due to erosion, abrasion and abfraction,
* Congenital anomalies,
* Cracked teeth were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2020-03-04 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Schiff Cold Air Sensitivity Scale Scores | Before treatment, immediately after treatment, 1 week, 1 month, 3 month and 6 month
  Average scores based on Schiff cold air sensitivity scale after evaporative air application. The Schiff score ranges from 0 to 3. Minimum value is 0, maximum value is 3. An increase in the score from 0 to 3 indicates an increase in sensitivity.
Visual Analog Scale(VAS) Scores | Before treatment, immediately after treatment, 1 week, 1 month, 3 month and 6 month
  Average scores based on Visual Analog Scale(VAS) after applying evaporative air. The VAS score ranges from 0 to 10. The minimum value is 0 and the maximum value is 10. A score of 0 is defined as "no pain" while a score of 10 is defined as "intolerable pain".
Dentin Hypersensitivity Experience Questionnaire (DHEQ) scores | Change from baseline quality of life at 6 months
  Data obtained after individuals complete the Dentin Hypersensitivity Experience Questionnaire. The decrease in the measured scores over time indicates that the quality of life has improved.

CONTACTS AND LOCATIONS:
Overall Officials: Behiye Esra Özdemir, Res. Assist., Principal Investigator — Kırıkkale University Faculty of Dentistry
Locations (1):
- Kırıkkale University Faculty of Dentistry, Department of Restorative Dentistry, Kırıkkale, Yahşihan/Kırıkkale, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: starting 6 months after publication
Access Criteria: Behiye Esra Özdemir

REFERENCES:
- [Result] Mason S, Burnett GR, Patel N, Patil A, Maclure R. Impact of toothpaste on oral health-related quality of life in people with dentine hypersensitivity. BMC Oral Health. 2019 Oct 22;19(1):226. doi: 10.1186/s12903-019-0919-x. PMID 31640741